CLINICAL TRIAL: NCT01409122
Title: A Phase 1, Placebo Controlled, Blinded, Multiple Dose Escalation Study of AIR001 (Sodium Nitrite Inhalation Solution) in Healthy Subjects, an Assessment of the Tolerability in Combination With Oral Sildenafil, and an Open-Label Study of Multiple Dose AIR001 in Patients With Pulmonary Arterial Hypertension
Brief Title: Safety, Tolerability, and PK Parameters of Sodium Nitrite Inhalation Solution in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aires Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AIR001-CS04
Record Dates: First submitted 2011-08-01; First posted 2011-08-04 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension
Keywords: vasodilator; nitric oxide; sodium nitrite; sildenafil; PDE-5; pulmonary hypertension; pulmonary arterial hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A Multiple Dose (Experimental): Ascending multiple dose administration (every 8 hours, [Q8H]) of AIR001 or placebo for 16 consecutive doses
  Interventions: Drug: 15 mg sodium nitrite inhalation solution; Drug: 90 mg sodium nitrite inhalation solution; Drug: 45 mg sodium nitrite inhalation solution; Drug: 120 mg sodium nitrite inhalation solution
- Part B Single Dose with Sildenafil (Experimental): Single escalating doses of AIR001 or placebo (Q8H, Day 4-6) administered in combination with steady-state sildenafil administration (Q8H, Days 1-6)
  Interventions: Drug: 25% MTD sodium nitrite inhalation solution
- Part C, administration of AIR001 to patients with PAH (Experimental): Four doses of AIR001 will be administered via nebulization to patients with PAH.
  Interventions: Drug: 90 mg sodium nitrite inhalation solution
- Part D, device crossover study (Experimental): PK, safety and tolerability of single doses of AIR001 administered in a randomized order with three different nebulizers.
  Interventions: Drug: 90 mg sodium nitrite inhalation solution

INTERVENTIONS:
Drug: 15 mg sodium nitrite inhalation solution — 15 mg sodium nitrite inhalation solution Q8H
  Arms: Part A Multiple Dose
Drug: 90 mg sodium nitrite inhalation solution — 90 mg sodium nitrite inhalation solution Q8H
  Arms: Part A Multiple Dose; Part C, administration of AIR001 to patients with PAH; Part D, device crossover study
Drug: 45 mg sodium nitrite inhalation solution — 45 mg sodium nitrite inhalation solution Q8H
  Arms: Part A Multiple Dose
Drug: 120 mg sodium nitrite inhalation solution — 120 mg sodium nitrite inhalation solution or placebo Q8H
  Arms: Part A Multiple Dose
Drug: 25% MTD sodium nitrite inhalation solution — Multiple oral doses of 20 mg sildenafil will be administered open-label Q8H to a single cohort of eight subjects on Days 1 to 6. A single dose of sodium nitrite inhalation solution equal to 25% of the maximum tolerated dose (MTD) identified in Part A (or placebo) will be administered on Day 4, a single dose equal to 50% of the MTD (or placebo) will be administered on Day 5, and a single dose equal to 100% of the MTD (or placebo) will be administered on Day 6.
  Arms: Part B Single Dose with Sildenafil

SUMMARY:
This is a four-part study of the safety, tolerability, and PK profile of sodium nitrite inhalation solution (AIR001) of ascending multiple doses (Part A) and of escalating doses with steady-state sildenafil (Part B) to healthy male and female subjects, as well as assessment of the safety and tolerability of multiple doses of AIR001 to patients with pulmonary arterial hypertension (part C) with a single dose PK study of AIR001 utilizing three different nebulizers (Part D).

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is an increase in the blood pressure (BP) in the small pulmonary vessels, arteries, veins or capillaries that results in progressive increases in right ventricular afterload, often leading to right ventricular failure and death. Pulmonary hypertension can result from a multitude of pathologies, including arterial etiologies, venous, chronic hypoxia related, thromboembolic, and other miscellaneous etiologies. In the recent Dana Point Classification, pulmonary arterial hypertension (PAH) was classified as Group 1. In Group 1 PAH, the pathologic lesion is localized to the small muscular pulmonary arteries, resulting in luminal narrowing and resistance to blood flow. Group 1 PAH includes idiopathic or sporadic PAH and heritable PAH which includes those with a family history of PAH. Associated PAH includes disease associated with connective tissue disease as well as PAH associated with congenital systemic to pulmonary shunts, portal hypertension, and human immunodeficiency virus (HIV) infection. Drug and toxin induced PAH is also in Group 1. Untreated, patients with PAH have an average life expectancy of 3 years, which declines to approximately 1 year if right heart failure is present.

Inhaled nitric oxide (NO) is a potent acute vasodilator. Its acute administration results in improved hemodynamics in the 10 to 15% of patients with PAH who demonstrate acute vasoreactivity. However, the usefulness of NO for chronic therapy is limited by the need for continuous inhalation. In patients who demonstrate vasoreactivity during an acute challenge with inhaled NO or a prostanoid challenge, therapy with calcium channel blockers has been demonstrated to result in improved symptoms and survival. In patients who do not demonstrate an acute vasodilator response, available therapies for PAH include prostanoids, endothelin receptor antagonists (ERA), and phosphodiesterase type-5 (PDE-5) inhibitors. However, the route and frequency of administration of the prostanoids, the hepatotoxicity of the ERAs, and concerns about the sustained efficacy of both the ERAs and PDE-5 inhibitors suggests that many patients with PAH could benefit from an effective therapy which offers ease of administration and a favorable toxicity profile.

Aires Pharmaceuticals, Inc. is developing a novel therapeutic, AIR001, for the treatment of PAH. The active ingredient in AIR001 is sodium nitrite, formulated in a buffered, pH-adjusted solution for nebulization. Preclinical data suggest that under the hypoxic, acidotic conditions present in the pulmonary hypertensive lung, inhaled sodium nitrite serves as a sustained release source of NO which will act as an acute pulmonary vasodilator. In addition, because decreased levels of NO have been shown to stimulate vascular remodeling, the increased NO resulting from nitrite inhalation is postulated to attenuate or reverse the pulmonary arterial remodeling process, resulting in both symptomatic improvement and pulmonary hemodynamic improvement in patients with PAH.

Preclinical experiments have shown that AIR001 by oral, IV, and inhalation routes of administration is effective in treating PAH induced by hypoxia or monocrotaline when administered as infrequently as once weekly at doses that generate plasma concentrations of approximately 1 to 10 uM and above. While the precise mechanism by which AIR001 exerts anti-hypertensive actions in PAH models remains to be elucidated, nitrite itself has been demonstrated to be metabolized to NO in animals and humans.

Single doses of AIR001 have been shown to be well tolerated in humans at dose levels that generate peak plasma concentrations (Cmax) in the target range established in preclinical models and no safety issues have been identified. AIR001 reduced PH induced by hypoxic gas inhalation in healthy volunteers at doses that are well tolerated. Preclinical and clinical data support further clinical investigation of inhaled AIR001 for the treatment of PAH. Before progressing to studies in patients with PAH, the safety and tolerability of multiple dose administration of AIR001 will be evaluated in Part A of the current study.

The PDE-5 inhibitor, sildenafil, is approved for use in patients with PAH and commonly used in the initial treatment for PAH. AIR001 is converted to NO, which increases cGMP dependent vasodilatation. Because PDE-5 inhibitors prevent the catabolism of cGMP by phosphodiesterase, it is possible that an exaggerated drug effect could be observed when AIR001 is administered to patients being treated with sildenafil. Therefore, combination safety and tolerability (in particular orthostatic effects) of escalating single doses of AIR001 will also be evaluated in combination with steady-state sildenafil in Part B of the study.

A cohort of patients with previously diagnosed PAH on stable background therapy will be assessed for safety and tolerability of multiple doses of AIR001 in Part C of the study.

Part D of the study will assess the PK, safety and tolerability of single dose AIR001 with each of three different nebulizers in a randomized crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Be informed of the nature of the study and is able to understand and has provided written informed voluntary consent
* Be healthy males or females, of any race, at least 18 years of age or the legal age of consent (whichever is greater) and less than 56 years of age at the time of the first dose of study drug (or sildenafil)
* Have a body mass index (BMI) >=18.0 and <32.0 kg/m2 and weigh at least 50 kg
* Be in good general health with no clinically relevant abnormalities based on the medical history, physical examination, clinical laboratory evaluations (hematology, clinical chemistry, urinalysis, methemoglobin), and 12-lead ECG that, in the opinion of the Investigator, would affect subject safety
* Agree to comply with the study procedures and restrictions

Exclusion Criteria:

* Any disease or condition that might affect drug absorption, metabolism, or excretion, or clinically significant cardiovascular, ocular, hematological, renal, hepatic, pulmonary, endocrine, gastrointestinal, immunological, dermatological, neurological, or psychiatric disease
* Clinically significant illness (including lower respiratory tract infection) or clinically significant surgery within 4 weeks before the administration of study drug (or sildenafil)
* Use of any commercially marketed mouthwash or oral rinse with agents other than tap water as well as tongue brushing or scraping from screening onwards through completion of study
* Currently a smoker or has a past history of smoking (of >10 pack years)
* History of bronchial asthma or sleep apnea
* Evidence of restrictive or obstructive lung disease (Forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity (FVC) <70%, FEV1 <70% predicted, and/or FVC <70% predicted)
* Family history of primary PH
* History of pulmonary embolism
* Evidence of supine hypertension or hypotension (systolic BP >180 mmHg or <90 mmHg and/or diastolic BP> 100 mmHg or <50 mmHg) pre-dose [NOTE: BP measurements may be repeated twice, at least 10 minutes apart]
* Orthostatic hypotension defined as a drop in systolic BP by >=20 mmHg or diastolic BP of >=10 mmHg at screening or predose or the development of significant postural symptoms (dizziness, lightheadedness, vertigo) when going from the supine to the standing position
* Personal or family history of congenital or acquired methemoglobinemia
* Personal or family history of RBC CYP B5 reductase deficiency
* Personal or family history or any evidence of hemoglobinopathy
* Known or suspected hypersensitivity or allergic reaction to sodium nitrite, sodium nitrate, or saccharin
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency or any contraindication to receiving methylene blue
* History of hypersensitivity or idiosyncratic reaction to drugs from multiple drug classes
* If female, is pregnant or breast feeding, or has a positive pregnancy test result pre-dose
* If a sexually active female, is not surgically sterile (defined as having had a hysterectomy, bilateral oophorectomy, or tubal ligation at least 6 months prior to screening) or post-menopausal (defined as amenorrhea for the past 2 years if <50 years of age or for the past 1 year if <=50 years or, if on hormone replacement therapy [HRT], documented follicle stimulating hormone [FSH] >30 IU/L before starting HRT), or does not agree to utilize two effective methods of contraception consistently and as intended from screening until at least 4 weeks after the last dose of study drug. Subjects must use a barrier method (diaphragm with intravaginal spermicide, cervical cap with intravaginal spermicide, or partner using condoms plus use of intravaginal spermicide) in combination with at least one of the following methods of contraception:

  1. systemic hormonal contraceptive (oral, implant, injection, or patch)
  2. intrauterine device
  3. or male partner who has undergone a vasectomy at least 6 months prior to screening.
* Unless approved by the Sponsor, chronic use of any systemic medications (with the exception of systemic hormonal contraceptives and vitamins taken at standard supplement doses); use of a drug therapy (including herbal preparations, e.g., St. John's wort) known to induce or inhibit hepatic drug metabolism within 30 days before the first dose of study drug (or sildenafil); use of prescription medication within 14 days before administration of study drug (or sildenafil) or over-the-counter [OTC] products (including natural products, vitamins) within 7 days before administration of study drug (or sildenafil). By exception, topical products without systemic absorption will be allowed. (NOTE: in particular, use of any PDE-5 inhibitor [e.g., sildenafil, tadalafil, vardenafil] is prohibited)
* Current history or evidence of drug abuse, history of regular alcohol consumption exceeding 21 drinks/week for men and 14 drinks/week for women (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of screening or a positive screen for substances of abuse or alcohol at screening or pre-dose
* Positive screen for hepatitis B surface antigen (HBsAg), hepatitis C antibody, or HIV antibody
* Receipt of an investigational product or device, or participation in a drug research study within a period of 30 days (or 5 half-lives of the drug, whichever is longer) before the first dose of study drug (sildenafil)
* Blood loss or blood donation of >550 mL within 90 days or plasma donation >500 mL within 14 days before administration of study drug (or sildenafil)
* Any food allergy, intolerance, restriction, or special diet that, in the opinion of the Investigator, should preclude the subject's participation in this study

Part B Only:

* Known or suspected hypersensitivity or allergic reaction to sildenafil or other therapeutics of similar chemical structure or any of the components of Revatio® tablets
* Any medical condition that constitutes a contraindication or risk to taking sildenafil, including a history of hereditary degenerative retinal disorders such as retinitis pigmentosa
* Ingestion of grapefruit or grapefruit juice within 72 hours before sildenafil administration

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ascending multiple dose AIR001 (Part A) | 16 doses administered Q8H over 5 days
  To evaluate the safety and tolerability of ascending multiple dose administration (every 8 hours, [Q8H]) of AIR001 for 16 consecutive doses
  * Adverse Events
  * 12 lead ECG
  * Vital Signs (change in supine BP, Pulse Rate and change in orthostatic BP)
  * Venous Methemoglobin
  * Spirometry
  * Percutaneous Saturation of Oxygen and Methemoglobin concentrations
  * Plasma cGMP
Safety and tolerability of single escalating doses of AIR001 with sildenafil (Part B) | 20 mg sildenafil Q8H for Days 1-6, single dose sodium nitrite inhalation solution over 10 min Days 4-6
  To evaluate the safety and tolerability of single escalating doses of AIR001 when administered in combination with steady-state sildenafil administration.
  * Adverse Events
  * 12 lead ECG
  * Vital Signs (change in supine BP, Pulse Rate and change in orthostatic BP)
  * Venous Methemoglobin
  * Spirometry
  * Percutaneous Saturation of Oxygen and Methemoglobin concentrations
  * Plasma cGMP
Composite PK for Plasma Nitrite and Nitrate(Part A) | following 1st dose of AIR001 on Day 1 and final dose on Day 6
  Cmax, tmax, AUC0-T, AUC0-inf, AUC%extrap, t½, CL/F, and Vz/F.
Composite PK for Plasma Nitrite and Nitrate in the presence of steady state Sildenafil(Part B) | Following the third dose of AIR001 on Day 5,6,7
  : Cmax, tmax, AUC0-T, AUC0-inf, AUC%extrap, t½,CL/F, and Vz/F.
Safety and tolerability of multiple doses of AIR001 administered to patients with PAH (PART C) | Multiple doses of sodium nitrite inhalation solution over 10 min for a total of 4 doses
  To evaluate the safety and tolerability of multiple doses of AIR001 when administered in combination with steady-state background PAH medications in patients with PAH.
  * Adverse Events
  * 12 lead ECG
  * Vital Signs (change in supine BP, Pulse Rate and change in orthostatic BP)
  * Venous Methemoglobin
  * Spirometry
  * Percutaneous Saturation of Oxygen and Methemoglobin concentrations
Safety and tolerability of single doses of AIR001 administered to healthy subjects with each of three different nebulizers (PART D) | Multiple doses of sodium nitrite inhalation solution over 10 min for a total of 4 doses
  To evaluate the safety and tolerability of single doses of AIR001 when administered in a randomized fashion with each of three different nebulizers in healthy volunteers.
  * Adverse Events
  * 12 lead ECG
  * Vital Signs (change in supine BP, Pulse Rate and change in orthostatic BP)
  * Venous Methemoglobin
  * Spirometry
  * Percutaneous Saturation of Oxygen and Methemoglobin concentrations
Composite PK for Plasma Nitrite and Nitrate(Part C) | following 1st dose of AIR001 on Day 1 and final dose on Day 2
  Cmax, tmax, AUC0-T, AUC0-inf, AUC%extrap, t½, CL/F, and Vz/F.
Composite PK for Plasma Nitrite and Nitrate(Part D) | following each dose of AIR001 with three different nebulizers
  Cmax, tmax, AUC0-T, AUC0-inf, AUC%extrap, t½, CL/F, and Vz/F.

CONTACTS AND LOCATIONS:
Overall Officials: Azra Hussaini, MD, Principal Investigator — PAREXEL International - Baltimore
Locations (1):
- PAREXEL International Early Phase Clinical Unit - Baltimore, Baltimore, Maryland, United States